CLINICAL TRIAL: NCT00004880
Title: A Phase I Pilot Trial of a Multi-Antigen Loaded Dendritic Cell Vaccine for the Treatment of Advanced Renal Cell Carcinoma
Brief Title: Vaccine Therapy in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067542; UCLA-9703025; NCI-G00-1675
Record Dates: First submitted 2000-03-07; First posted 2004-05-20 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: dendritic cell vaccine therapy
Procedure: conventional surgery

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety of multiantigen loaded dendritic cells (DC) vaccine in patients with advanced renal cell carcinoma. II. Evaluate the immunologic response to this regimen in this patient population. III. Evaluate the clinical response to this regimen in this patient population.

OUTLINE: This is a sequential cohort study. All patients undergo total nephrectomy to harvest primary tumor for vaccine preparation. Patients without primary tumor undergo surgical resection of the accessible metastatic site for vaccine preparation. Patients are assigned to 1 of 4 treatment arms. Arm I: Patients receive vaccination with irradiated autologous tumor lysate (TuLy) intradermally (ID) on day 0 followed by vaccination with multiantigen liposome loaded dendritic cells (DC) ID on days 7, 14, and 21. Arm II: Patients receive vaccinations as in arm I, except DC are pulsed with tumor cells. Arm III: Patients receive vaccination with irradiated autologous tumor lysate (TuLy) IV on day 0 followed by vaccination with multiantigen liposome loaded DC IV on days 7, 14, and 21. Arm IV: Patients receive vaccinations as in arm III, except DC are treated as in arm II. Patients are followed on days 28, 42, 70, and 112.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic renal cell carcinoma Evaluable or bidimensionally measurable disease with primary renal tumor in place or surgically accessible metastatic site greater than 2 x 2 cm
* Over 18
* ECOG 0-1
* Hematopoietic:

  * Hemoglobin at least 10 g/dL (not transfusion dependent)
  * Platelet count at least 75,000/mm3
  * WBC greater than 3,000/mm3
* Hepatic: SGOT/SGPT no greater than 5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN
* PT/PTT no greater than 1.5 times ULN
* Bilirubin no greater than 2.5 mg/dL
* Renal: Creatinine no greater than 2.0 g/dL
* Hepatitis B surface antigen negative
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 4 weeks since prior immunotherapy
* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior radiotherapy
* At least 14 days since prior acute therapy for infection

Exclusion Criteria:

* uncontrolled CNS metastasis
* ischemic heart disease that precludes surgery
* pulmonary condition that precludes surgery
* other underlying condition or allergy that would preclude study
* acute viral, bacterial, or fungal infection requiring therapy HIV negative
* pregnant or nursing
* other acute medical problems that would preclude study
* concurrent corticosteroids (oral, topical, inhaled)
* prior organ allografts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1997-06; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Gitlitz, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States